CLINICAL TRIAL: NCT05730361
Title: Phase Ib Clinical Study on the Safety, the Tolerability, the Pharmacokinetics and the Efficacy of ScTIL Injection (Gene Modified Tumor Infiltrating Lymphocytes) Alone and in Combination With B Lymphocyte Adjuvant in the Treatment of Digestive System Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director of Department of Gastroenterology and oncology, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ScTIL-B-009-2022
Record Dates: First submitted 2023-02-07; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-11

CONDITIONS: Digestive System Malignant Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ScTIL injection (Experimental): This trial is designed single arm. All the subjects enrolled will receive the experimental intervention: ScTIL210 injection alone or with B lymphocytes adjuvant.
  Interventions: Biological: ScTIL injection; Biological: ScTIL injection and B lymphocytes adjuvant

INTERVENTIONS:
Biological: ScTIL injection — Peripheral blood mononuclear cells (PBMCs) obtained via apheresis are used for cell preparation. PD-1 positive T cells are isolated from PBMCs, are transduced with lentivirus loaded with "enhanced receptor" and "superamplification factor", and cell number are amplified. The obtained ScTIL is used for one-time intravenous infusion.
Biological: ScTIL injection and B lymphocytes adjuvant — B lymphocyte are also isolated from PBMCs. If the percentage of subject's B lymphocyte in total lymphocytes is > 5%, the autologous B lymphocyte adjuvant will be prepared. If this percentage is ≤ 5%, PBMCs will be collected from haploidentical donor of the subject via apheresis, and B lymphocyte will be isolated for preparation of allogeneic B lymphocyte adjuvant.

SUMMARY:
This is an open-lable, single-arm, single-dose escalation and multiple-dose extention clinical study of cell therapy designed to observe and evaluate the tolerance, the pharmacokinetic characteristics, the safety and the efficacy of ScTIL210 injection alone and in combination with B lymphocytes adjuvant in the treatment of digestive system malignant solid tumors.

DETAILED DESCRIPTION:
This study consists of two phases: the first phase will be the dose exploration phase (Phase I), followed by the dose extension phase (Phase II).

In phase I, 3 subjects are enrolled for 1st treatment group, starting with single dose of ScTIL injection of 5x10^9 alone. If there is no dose limiting toxicity (DLT) observed, 3 subjects are enrolled into treatment groups successively in sequential order of: 1) Group 2: ScTIL1.5x10^10 alone; 2) Group 3: ScTIL 5x10^9 plus B lymphocytes adjuvant 5x10^9; and 3) Gorup 4: ScTIL1.5x10^10 plus B lymphocytes adjuvant 1.5x10^10. Preconditioning chemotherapy will be performed to subjects of 3rd and 4th treatment group. Fludarabine 25mg/m2/day and cyclophosphamide 250mg/m2/day will be intravenously administered at 5 and 4 days (Day -5 and Day -4) before reinfusion of ScTIL and B lymphocyte adjuvant at Day 0.

After the completion of ScTIL reinfusion for first subject of the 1st dose group, the subject will be observed for no less than one week. If no serious toxic and adverse events occurres, ScTIL reinfusion for the second and third subjects will be performed. If no DLT occurres by the 14th days after completion of reinfusion for the 3rd subject, The study will move to the next treatment group. If 1/3 of enrolled subjects have DLT, another 3 subjects will be enrolled. In any of the dose groups, if ≤1/6 subjects have DLT, subject enrollment for the next treatment group will start. If DLT occurs in ≥2/6 of subjects, the number of subjects in the previous dose group shall be reviewed. If there were only 3 subjects, 3 more subjects will be enrolled. If DLT occurs in ≤1/6 subjects, the dose will be defined as the maximum tolerable dose (MTD), and the dose escalation phase of the study will be completed. If DLT occurs in ≥2/6 subjects in the first dose group, a dose reduction exploration will be performed or the study will be terminated upon decision made by the Safety Committee. A independent third party safety audit committee (consists of no clinical study participants) will conduct safety audit 14 days after the first ScTIL reinfusion of the third subject of the 1st treatment group.

In phase II, If no dose limiting toxicity event occurred after the completion of treatment in each of the 4 groups. Researcher will decide to select 2-4 dose groups for dose extention study and will enroll 5-10 subjects for each group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75, regardless of gender;
2. Expected survival time > 3 months;
3. Patients with digestive system malignant solid tumors (esophageal cancer, gastric cancer, pancreatic cancer, colorectal cancer, etc.) who have failed the standard treatment confirmed by histology or cytology, or have disease progression after multi-line treatments, or are currently not suitable for standard treatment;
4. PD-1 positive T cells in peripheral blood accounted for≥ 18% of total T lymphocytes;
5. Voluntarily accept the use of peripheral blood cell apheresis to obtain cells for the preparation of ScTIL cells; On the premise of informed consent, haploidentical cell donors (lineal blood relatives: parents, children, brothers and sisters) are sampled and detected for HLA matching, infectious disease index, blood routine examination, bleeding, and coagulation indicators, followed by collection of peripheral blood mononuclear cells (PBMCs ≥ 3x10^9) via apheresis of the cell donors to prepare allogeneic B lymphocyte adjuvant;
6. According to RECIST version 1.1, there is at least one measurable tumor focus. The measurable tumor focus is defined as the longest diameter ≥ 10mm and the CT scanning thickness does not exceed 5.0mm. For lymph node lesions, the short diameter ≥ 15mm;
7. The Eastern Cooperative Oncology Group (ECOG) physical condition score is 0 to 1;
8. Sufficient bone marrow and organ functions:

   1. Hematology: neutrophils is equal to or higher than 1.5×10^9/L, platelets is equal to or higher than 75×10^9/L, hemoglobin is equal to or higher than 90g/L; total lymphocytes is equal to or higher than 50% of the lower limit of normal range;
   2. Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are both eqal to or lower than 3 times the upper limit of normal range (ULN) (if intrahepatic bile duct cancer exists, equal to lower than 5 times of ULN); total bilirubin (TBIL) is equal to or lower than 2 times of ULN;
   3. Kidney function: Creatinine (Cr) is equal to or lower than 1.5 times of ULN;
   4. Coagulation function: prothrombin time (PT) is equal to or shorter than 1.5 times of ULN or activated partial prothrombin time (APTT) is equal to or shorter than1.5 times of ULN;
   5. Urine protein concentration is equal to or lower than ≤ 1+, with no edema.
   6. Albumin is equal to or higher than 3.0g/dl.
9. Qualified patients with fertility (male and female) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence, etc.) with their partners during the trial and at least 90 days after the last medication; The blood or urine pregnancy test within 7 days before the first use of the study drug in women of childbearing age (see Appendix 8 for the definition) must be negative;
10. Be able to understand the study and to voluntarily sign the written informed consent.

Exclusion Criteria:

1. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence shows that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, so it is not suitable to be included in the study according to the judgment of the researcher;
2. Received systemic chemotherapy, radiotherapy, immunotherapy, anti-tumor bioactive traditional Chinese medicine and other anti-tumor treatments within 2 weeks before apheresis, except for the following:

   1. Nitrosourea or mitomycin C within 6 weeks before harvest;
   2. Oral fluorouracil and small molecule targeted drugs were taken 1 week before single harvest;
3. Received systemic glucocorticoid (prednisone > 10mg/day or equivalent dose of similar drugs) or other immunosuppressant treatment within 2 weeks before apheresis; Except for the following cases: Intermittent use of local, eye, intra-articular, intranasal and inhaled glucocorticoids; Short term use of glucocorticoids for preventive treatment (e.g. prevention of contrast agent allergy);
4. Within 4 weeks before apheresis:

   1. Have received other unlisted clinical research drugs or treatments;
   2. Having undergone major organ surgery (excluding puncture biopsy) or significant trauma, or requires scheduled hospitalization during the trial period;
   3. Used live attenuated vaccine;
5. There was active infection within 1 week before apheresis, and systemic anti-infection treatment was currently required;
6. Patients receiving PD-L1 mAb within 3 months before apheresis (Including but not limited to atilizumab and duvalizumab);
7. Imaging findings suggests the presence of progressive pulmonary autoimmune interstitial or alveolar inflammation;
8. Had received immunotherapy and had ≥ grade 3 IrAE (except hypothyroidism);
9. The adverse reaction of previous anti-tumor treatment has not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except for the toxicity without safety risk judged by researchers such as hair loss);
10. Patients with active or had autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.); Except for patients with clinically stable autoimmune thyroid disease and well controlled type I diabetes;
11. Have a history of immunodeficiency, including HIV antibody test positive;
12. Hepatitis B (immunological test results do not exclude infectivity) and/or hepatitis B DNA titer is higher than the lower limit of the detection value of the research center; And/or hepatitis C (anti HCV antibody positive); And/or treponema pallidum antibody positive;
13. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    1. There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, ⅱ - ⅲ degree atrioventricular blockade, etc;
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events ≥ grade 3 occurred within 6 months before the cell reinfusion;
    3. New York Heart Association (NYHA) cardiac function rating ≥ class II or left ventricular ejection fraction (LVEF) < 50%, or structural heart disease with high risk judged by other researchers;
    4. Clinically uncontrollable hypertension;
14. Serous cavity effusion beyond clinical control is not suitable for the group according to the judgment of the researcher;
15. Known alcohol or drug dependence;
16. Mental disorders or poor compliance;
17. Pregnant or lactating women;
18. The researcher believes that the subject has a history of other serious systemic diseases or is not suitable to participate in this clinical study due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 weeks after single dose of cell reinfusion
  Including cases of PR and of CR

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 12 weeks after single dose of cell reinfusion
  The number of cases with remission and stable lesions after treatment accounted for the total number of evaluable cases
Duration of Response (DOR) | 12 weeks after single dose of cell reinfusion
  Time from complete remission (CR) or partial remission (PR) to disease progression (PD), death or last tumor evaluation
Progression-Free Survival (PFS) | 12 weeks after single dose of cell reinfusion
  From the beginning of cell therapy to the time of the first disease progression or death due to any cause
Overall survival (OS) | Single dose of cell reinfusion to death
  Time from cell reinfusion to death due to any cause
Adverse events (AEs) | 24 weeks after single dose of cell reinfusion
  According to National Cancer Institute Common Terminology Criteria for Adverse Events V5.0(CTCAE V5.0)
Detection of Lentivirus Copy Number | 12 weeks after single dose of cell reinfusion
  Dynamic changes of carrier gene copy number in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Prof. Dr., Principal Investigator — Locations: Beijing University Cancer Hospital, Beijing, China, 100142